CLINICAL TRIAL: NCT02500719
Title: Real-time Functional MRI and Neurofeedback of Brain Networks Mediating Trauma Memory Recall in PTSD
Brief Title: Real-time fMRI and Neurofeedback of Brain Networks Mediating Trauma Memory Recall in PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 203600
Record Dates: First submitted 2015-07-07; First posted 2015-07-16 (Estimated); Results first posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-04

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Post-Traumatic Stress Disorder; Neurofeedback; fMRI; Skin Conductance Response
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Healthy Participants (Experimental): A group of healthy participants will be enrolled first in the pilot phase of the study. This phase allows for the refinement (prior to the implementing in our PTSD participant group) the application of our support vector machine based real-time functional magnetic resonance imaging (rt-fMRI) algorithm, which evaluates brain networks thought to mediate emotional arousal and presents them (in real time) to subjects to aide in volitional manipulation of arousal.
  Interventions: Device: Computational Model - Real-time Support Vector Machine
- PTSD Participants (Experimental): A group of participants with symptoms of PTSD will be enrolled in the implementation phase of the study. This phase allows for the evaluation of rt-fMRI guidance of brain networks thought to mediate emotional arousal, specifically whether participants can learn volitional control of these networks.
  Interventions: Device: Computational Model - Real-time Support Vector Machine

INTERVENTIONS:
Device: Computational Model - Real-time Support Vector Machine — A support vector machine algorithm will be applied in real-time to fMRI data to identify distributed patterns of co-activated brain regions that specifically encode high emotional arousal (i.e,. high SCR) to the stress/trauma memory (note, this is equivalent to predictions of fitted Q-iteration in which the all actions are specified as zero, reward is equal to the support vector machine predicted arousal, and the discount factor of 0). The resulting idiosyncratic brain map would inform the neurofeedback phase in the next stage of fMRI data collection. This approach will first be piloted in the healthy participant group, then implemented in the PTSD participant group.
  Other Names: Machine Learning Algorithm; Real-time Neurofeedback

SUMMARY:
The purpose of the current study is to develop a better understanding of the brain mechanisms involved in psychological treatments for posttraumatic stress disorder (PTSD). This project will build on past research using script-driven imagery in our lab by investigating brain activity in areas activated during exposure to trauma-related cues. This project will also develop new knowledge concerning volitional control of those areas. The ultimate goal of this study is a better understanding of whether volitional control of these brain areas will improve therapeutic outcomes. This process will first be piloted in a sample of healthy controls. This will allow investigators to refine the methodology prior to recruiting a sample with PTSD.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is characterized by intense emotional distress upon exposure to trauma reminders and avoidance of people and places that can trigger the trauma memory. Neurocircuitry models of PTSD that seek to explain symptoms of heightened emotional reactivity, hypervigilance for threat, and avoidance suggest abnormal activity of neural regions involved in emotional reactivity (e.g., amygdala) and cognitive control of emotional responding (e.g., ventral medial prefrontal cortex, anterior cingulate cortex). While knowledge exists about neurobiological abnormalities associated with PTSD, these data are cross-sectional in nature and ignore individual differences in both neural encoding and subjective aspects of the trauma itself (e.g., whether it elicits fear vs guilt vs disgust). Additionally, the manner by which existing psychological treatments alter these neural mechanisms mediating core PTSD symptoms is unknown. This is problematic, given that state-of-the-art treatment for PTSD is only effective ~60% of the time.

Here, the investigator proposes to utilize a novel computational modeling approach combined with state-of-the-art functional magnetic resonance imaging (fMRI)-based neurofeedback to directly identify and modulate the idiosyncratic neural network encoding the trauma memory. Successful pursuit of these aims would 1) provide scientific support for the hypothesis that a distributed network including the amygdala, hippocampus, medial prefrontal cortex (PFC), lateral PFC, and anterior insula mediates emotional responding upon trauma memory recall, and 2) provide proof-of-concept evidence that neurofeedback modulation of this network can boost existing therapy efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 21-50
* Medically healthy

Exclusion Criteria:

* Claustrophobia, or the inability to lie still in a confined space
* Major medical disorders (e.g., HIV, cancer)
* Magnetic metallic implants (such as screws, pins, shrapnel remnants, aneurysm clips, artificial heart valves, inner ear (cochlear) implants, artificial joints, and vascular stents)
* Electronic or magnetic implants, such as pacemakers
* Permanent makeup or tattoos with metallic dyes
* Currently pregnant
* A self-reported history of loss of consciousness (greater than 10 minutes)
* Physical disabilities that prohibit task performance (such as blindness or deafness)
* Psychotic disorders (e.g., schizophrenia)
* Any other condition that the investigator believes might put the participant at risk

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-15 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Bush, PhD., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants: A group of healthy participants will be enrolled first in the pilot phase of the study. This phase allows for the refinement (prior to the implementing in our PTSD participant group) the application of our support vector machine based real-time functional magnetic resonance imaging (rt-fMRI) algorithm, which evaluates brain networks thought to mediate emotional arousal and presents them (in real time) to subjects to aide in volitional manipulation of arousal.
  Computational Model - Real-time Support Vector Machine: A support vector machine algorithm will be applied in real-time to fMRI data to identify distributed patterns of co-activated brain regions that specifically encode high emotional arousal (i.e,. high SCR) to the stress/trauma memory. The resulting idiosyncratic brain map would inform the neurofeedback phase in the next stage of fMRI data collection. This approach will first be piloted in the healthy participant group, then implemented in the PTSD participant group.
- PTSD Participants: A group of participants with symptoms of PTSD will be enrolled in the implementation phase of the study. This phase allows for the evaluation of rt-fMRI guidance of brain networks thought to mediate emotional arousal, specifically whether participants can learn volitional control of these networks.
  Computational Model - Real-time Support Vector Machine: A support vector machine algorithm will be applied in real-time to fMRI data to identify distributed patterns of co-activated brain regions that specifically encode high emotional arousal (i.e,. high SCR) to the stress/trauma memory. The resulting idiosyncratic brain map would inform the neurofeedback phase in the next stage of fMRI data collection. This approach will first be piloted in the healthy participant group, then implemented in the PTSD participant group.
Period: Overall Study
Arm/Group | Healthy Participants | PTSD Participants
Started | 14 | 16
Completed | 11 | 9
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 2 | 3
Not completed — Trauma history | 1 | 0
Not completed — MRI data found to be unusable during analysis | 0 | 1
Not completed — Did not meet criteria for PTSD | 0 | 1
Not completed — Claustrophobia | 0 | 1
Not completed — History of head trauma | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | PTSD Participants | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Screen failure: Trauma history reported and subject age not recorded.
  years
    number analyzed (Participants) | 13 | 16 | 29
    (all) | 31.23 (8.30) | 32.5 (9.63) | 31.93 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 16 | 30
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 14 | 15 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 12 | 12 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Patient Emotional Response to Volitional Engagement and Disengagement of Emotional Arousal as Measured Using Support Vector Machine Decodings When the Decoding is Provided as Real-time Neurofeedback Guidance or Not.
Description: Support vector machine decodings of functional MRI data acquired during volitional engagement or disengagement of emotional arousal. Each decoding represents the Euclidean distance and direction (either positive or negative) of the functional MRI data volume with respect to the patient's support vector machine decision hyperplane. Positive distances denote engagement of emotional arousal and negative distances denote disengagement of emotion arousal. Distance represents the magnitude of volitional engagement or disengagement. Decodings can either be provided to patients as real-time neurofeedback (via visual representation of the distance) or hidden from view. When hidden, the visual representation of neurofeedback remains stationary.
Time Frame: Real-time within the measurement of functional MRI (within 10 seconds of functional MRI volume acquisition and reconstruction)
Population: Completing subjects.
Measure: Mean (Standard Deviation); unit: Standard score (decodings)
Units Other Than Participants: Decodings
Arm/Group | Healthy Participants | PTSD Participants
Number analyzed (Participants) | 11 | 9
Number analyzed (Decodings) | 875 | 800
Standard score (decodings)
  Volitional Engagement of Arousal Achieved without Real-time Neurofeedback Guidance. | -.2104 (.7311) | .4659 (1.194)
  Volitional Disengagement of Arousal Achieved without Real-time Neurofeedback Guidance. | -.2952 (.8211) | .0080 (.9234)
  Volitional Engagement of Arousal Achieved with Real-time Neurofeedback Guidance. | -.0257 (.7762) | .5244 (1.319)
  Volitional Disengagement of Arousal Achieved with Real-time Neurofeedback Guidance. | -.3186 (.8262) | -.0654 (.9453)
Statistical Analysis 1: Comparison: PTSD Participants; This test is to determine if the difference between engagement and disengagement of emotional arousal is increased by real-time neurofeedback guidance in PTSD participants; Test type: Superiority; p = .029, t-test, 1 sided; Mean Difference (Net) = .1319

ADVERSE EVENTS:
Time Frame: 3 hours
Arm/Group | Healthy Participants | PTSD Participants
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT02500719/Prot_SAP_000.pdf